CLINICAL TRIAL: NCT03397927
Title: The Improved Ballet Shoe: a Study on the Effect of an Orthosis on Pain During Dancing on Pointe Shoes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No response to EC questions were given
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 133057
Record Dates: First submitted 2014-01-23; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2014-01

CONDITIONS: Ballet Dancers
Keywords: ballet shoe; orthosis; pain
MeSH Terms: conditions — Pain | interventions — Orthotic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- orthosis (Experimental)
  Interventions: Device: orthosis

INTERVENTIONS:
Device: orthosis

SUMMARY:
An orthosis in the ballet shoe to see if pain reduction during dancing on pointes will decrease.

One group of pre-preprofessional ballet dancers will receive an orthosis and will train during four weeks with it. The other group without a orthosis will be the control group.

ELIGIBILITY:
Inclusion Criteria:

* girls on preprofessional ballet schools with a minimum of 30 minutes professional training a week;
* 12 to 18 years old
* pain during dancing on pointes

Exclusion Criteria:

* experience with wearing a orthosis in their ballet shoe

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
VAS-score | four weeks

SECONDARY OUTCOMES:
lower extremities muscle ratio | four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands